CLINICAL TRIAL: NCT00778453
Title: Relative Effects and Predictive Models of Contemporary Upper Limb Training Programs in Stroke Patients Delivered in Hospital-based and Home-based Settings
Brief Title: Relative Effects and Predictive Models of Contemporary Upper Limb Training Programs in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Ching-yi Wu, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSC97-2314-B-182-004-MY3; 96-1754B (Other: Institutional Review Board / Chang Gung Memorial Hospital)
Record Dates: First submitted 2008-10-05; First posted 2008-10-23 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Cerebrovascular Accidents
Keywords: stroke rehabilitation; kinematic analysis; upper extremity training; predictors
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Hospital-based mCIT (Experimental): Hospital-based modified constraint-induced therapy(mCIT)
  Interventions: Other: Hospital-based mCIT
- Hospital-based BIT (Experimental): Hospital-based bilateral isokinematic training (BIT)
  Interventions: Other: Hospital-based BIT
- Hospital-based TR (Experimental): Hospital-based traditional rehabilitation (TR)
  Interventions: Other: Hospital-based TR
- Home-based BAT (Experimental): Home-based bilateral arm training(BAT)
  Interventions: Other: Home-based BAT
- Home-based TR (Experimental): Home-based traditional rehabilitation (TR)
  Interventions: Other: Home-based TR
- Home-based mCIT (Experimental): Home-based modified constraint-induced therapy (mCIT)
  Interventions: Other: Home-based mCIT

INTERVENTIONS:
Other: Hospital-based mCIT — restraint of the unaffected arm and practice of the affected arm
  Other Names: Hospital-based modified constraint-induced therapy(mCIT)
  Arms: Hospital-based mCIT
Other: Hospital-based BIT — bilateral symmetric, repetitive arm training
  Other Names: Hospital-based bilateral isokinematic training (BIT)
  Arms: Hospital-based BIT
Other: Hospital-based TR — hospital-based traditional rehabilitation : OT or PT or therapist-based training
  Other Names: Hospital-based traditional rehabilitation (TR)
  Arms: Hospital-based TR
Other: Home-based mCIT — restraint of the unaffected arm and practices of the affected arm
  Other Names: Home-based modified constraint-induced therapy (mCIT)
  Arms: Home-based mCIT
Other: Home-based BAT — bilateral symmetric, repetitive arm training
  Other Names: Home-based bilateral arm training (BAT)
  Arms: Home-based BAT
Other: Home-based TR — home-based traditional rehabilitation:OT or PT or therapist-based training
  Other Names: Home-based traditional rehabilitation (TR)
  Arms: Home-based TR

SUMMARY:
The findings of this study will advance movement reorganization mechanism underlying treatment approaches and clinical intervention techniques. These findings may inform rehabilitation professionals about which treatment approach is superior to another one in certain aspect of outcome and who can benefit most from certain treatment approach. Accordingly, the results of this project may help us move quickly to design and develop efficient and effective rehabilitation programs for individualized patients.

DETAILED DESCRIPTION:
The first purpose is to investigate the relative effects of modified constraint-induced therapy (mCIT) vs. bilateral isokinematic training (BIT) vs. traditional or therapist-based training (TR) on movement reorganization, motor performance, functional ability, and quality of life (QoL) immediately and six months later after treatment delivered at hospitals. Movement reorganization will be evaluated by kinematic instrument. Motor performance, functional ability, and QoL will be assessed using clinical assessment tools. By the same token, we also investigate the relative effects of these two approaches delivered at home. The second purpose is to study whether home-based mCIT is efficacious in various aspects of outcomes described above immediately and six months later following treatment, compared to home-based TR, and hospital-based mCIT and TR.We also study the same question regarding home-based BIT efficacy. The third purpose is to establish predictive models to predict functional and QoL outcomes immediately and six months later following mCIT and BIT.

ELIGIBILITY:
Inclusion Criteria:

* the onset duration more than 6 months
* Brunnstrom stage III above for the proximal part and distal part of UL
* no serious cognitive deficits
* no balance problems sufficient to compromise safety when wearing the project's constraint device
* no excessive spasticity in any of the joints of the affected UL exclusion criteria:
* a score of less than 24 on the Mini Mental State Exam

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
kinematic analysis | 2008-2011

SECONDARY OUTCOMES:
clinical measures | 2008-2011

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Department of Occupational Therapy, Chang Gung Univ
Locations (1):
- Chang Gung Memorial Hospital, Kwei-shan, Toayuan, Taiwan

REFERENCES:
- [Derived] Lin KC, Chuang LL, Wu CY, Hsieh YW, Chang WY. Responsiveness and validity of three dexterous function measures in stroke rehabilitation. J Rehabil Res Dev. 2010;47(6):563-71. doi: 10.1682/jrrd.2009.09.0155. PMID 20848369